CLINICAL TRIAL: NCT03602937
Title: A Study to Evaluate the Acceptability and Nutritional Suitability of Renastep, a Food for Special Medical Purposes (FSMP) for Use in the Dietary Management of Patients From 3-18 Years of Age With Chronic Kidney Disease (CKD)
Brief Title: Evaluation of Renastep
Acronym: Renastep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitaflo International, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCT-RENS-2017-11-07
Record Dates: First submitted 2018-04-23; First posted 2018-07-27 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Chronic Kidney Diseases; Renal Disease
Keywords: Acceptability; Renal; CKD; Kidney; Vitaflo; High energy, low volume; Low potassium; Low phosphorus; Low vitamin A
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases

STUDY DESIGN:
Intervention Model Description: Open label prospective acceptability study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Renastep (Experimental): All participants to incorporate Renastep into their usual dietary regime.
  Interventions: Dietary Supplement: Renastep

INTERVENTIONS:
Dietary Supplement: Renastep — Renastep is a ready-to-use, high energy, low volume liquid renal specific feed that can be administered enterally via tube or oral consumption.

SUMMARY:
Evaluation of Renastep is a 28-day long, prospective nutritional study that will recruit 15 patients aged between 3 and 18 years of age with Chronic Kidney Disease. Participants will incorporate Renastep into their renal specific diet, during which time they will record gastrointestinal symptoms, adherence to recommended intakes and thoughts on its palatability. A Baseline CRF completed by the Investigator at the start of the trial will record demographic information, GI history and the most recent renal bio-marker results. Bio-marker results recorded as part of routine care over the course of the study will be captured in the End of Study CRF.

The study is designed to generate acceptability data that will be used to support an application to the Advisory Committee on Borderline Substances for Renastep to be reimbursable on prescription within the NHS.

DETAILED DESCRIPTION:
Renastep is designed for use in the dietary management of kidney disease between 3 and 18 years of age. It is a high-energy liquid feed containing protein, carbohydrate, fat, vitamins, minerals, trace elements and DHA. It contains low levels of potassium, phosphorus, calcium, chloride and vitamin A compared with a standard paediatric enteral feed.

Vitaflo (International) Ltd has developed Renastep following a request from the Paediatric Renal Interest Nutrition Group (PRING). They requested a low potassium and phosphate, high energy liquid feed for the dietary management of children with kidney disease that can be used as a sip feed or as a part of a modular tube feed.

There is currently no product designed specifically for use in this age group. Current dietetic practice involves either prescribing a powdered infant formula, in variable concentrations, or manipulating an adult renal sip feed to construct a modular feed, meeting the particular individual requirements of a paediatric patient with chronic kidney disease. This can be time consuming, complicated, can frequently involve preparation error leading to over or underconcentration of key nutrients, and increases the risk of microbial contamination. As Renastep is a ready to use product designed specifically for children with kidney disease, it can be expected that it will be more easily incorporated into the dietary management of the patient than the current options available. This has also been requested by the children and their families. Renastep could replace unsafe current practices that are the only option available to clinicians.

In order for Renastep to be prescribed within the NHS, it must first be subject to an application to the Advisory Committee on Borderline Substances (ACBS). The ACBS require data on the product's acceptability, in terms of gastrointestinal tolerance, palatability and participants' adherence to recommended intakes. The ACBS require such acceptability studies to be conducted in at least 15 patients for whom the product is designed. This stipulation is the reason for conducting the trial within patients aged 3 - 18 years of age with Chronic Kidney Disease.

The study will last for 28 days. Participants will self-report study data in Daily Diary forms that include 7 days of gastrointestinal data, daily records of how much of the product has been taken compared to the amount prescribed and a final evaluation of the product's palatability. The investigator will complete a Baseline CRF at the first visit to record demographic information, GI history and the most recent urea, phosphorus and potassium results. This will be supplemented by an End of Study CRF which will record urea, phosphorus and potassium results recorded during the trial period as part of usual clinical care. Information relating to gastrointestinal tolerance of Renastep over the 28-day study period will also be recorded by the Investigator in the End of Study CRF.

All study data will be anonymised and reviewed by the local investigator prior to it being forwarded to the sponsor, Vitaflo (International) Ltd.

ELIGIBILITY:
Inclusion Criteria:

i) Diagnosis of Chronic Kidney Disease.

ii) Aged between 3 and 18 years.

iii) Has a requirement for a restricted potassium and/or restricted phosphorus diet.

iv) Has a requirement for nutrition support.

v) Freely given, written, informed consent from patient or parent/guardian.

vi) Freely given, written assent (if appropriate).

Exclusion Criteria:

i) Inability to comply with the study protocol, in the opinion of the investigator.

ii) Aged under 3 years or over 18 years.

iii) Use of additional enteral feeds during the study period, unless clinically indicated and prescribed by the investigator (must be recorded in patient case record file).

iv) Women who are pregnant / breastfeeding at the start of the study or planning to become pregnant during the study period.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Patients' compliance with recommended intakes of Renastep. | Days 1 - 28.
  Actual intake of the product will be compared with recommended intake. Participant to record how much of the product they took on each of the study days in a daily study dairy.
Patients' gastrointestinal tolerance of Renastep. | Days 1 - 7.
  Participant to record any gastrointestinal symptoms experienced in a daily study diary.
Patients' thoughts on Renastep's palatability | Day 28.
  Participants will rate Renastep's appearance, smell, taste, aftertaste, texture and presentation on a 5-point Likert scale at the end of their time on the study.
Patients' thoughts on Renastep's ease of use | Day 28.
  Participants will rate Renastep's ease of use on a 5-point likert scale at the end of their time on the study.
Nutritional suitability | Days 0 - 28
  The product's nutritional suitability for use in a renal specific diet will be measured. The investigator will record the participant's most recent urea, phosphorus and potassium results (all mmo/L) taken as part of routine care prior to the intervention period beginning and all available results recorded as part of routine care over the course of the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Anderson, Study Director — University Hospital Southampton NHS Foundation Trust; Alison Holmes, Principal Investigator — Alder Hey Children's NHS Foundation Trust; Sara Janes, Principal Investigator — Birmingham Women's and Children's NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - Southampton Children's Hospital, Southampton, Hampshire
  - Alder Hey Children's Hospital, Liverpool, Merseyside
  - Birmingham Children's Hospital, Birmingham, West Midlands

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.